CLINICAL TRIAL: NCT01341600
Title: Clopidogrel Pharmacogenetics Bench to Bedside - A Practical Application
Brief Title: Clopidogrel Pharmacogenetics (PGX) Bench to Bedside
Acronym: PGXB2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Cancer Institute (NCI) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alan Shuldiner, Professor of Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP-00044487; U01GM074518 (NIH); U01HL105198 (NIH); 128475 (Other Grant/Funding Number: NIH); ZICSC006536 (NIH); ZICSC006537 (NIH)
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Metabolism of Clopidogrel
Keywords: Clopidogrel; Pharmacogenetics; Platelets; Healthy Subjects
MeSH Terms: interventions — Clopidogrel; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Clopidogrel in poor metabolizers (Experimental): Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI) will be recruited. We will select 6 poor metabolizers (PM) to clopidogrel 75 mg from participants who previously received 75 mg clopidogrel as part of another NIH sponsored clinical trial entitled, "Pharmacogenetics of Anti-platelet Intervention" (PAPI) Study (NCT 00799396). Over a 6 week period participants will be given: 75 mg of clopidogrel for 8 days, at least 1 week washout, 150 mg of clopidogrel for eight days, at least 1 week washout, 300 mg of clopidogrel for eight days.
  Interventions: Drug: Clopidogrel
- Clopidogrel in intermediate metabolizers (Experimental): Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI) will be recruited. We will select 6 intermediate metabolizers (IM) to clopidogrel 75 mg from participants who previously received 75 mg clopidogrel as part of another NIH sponsored clinical trial entitled, "Pharmacogenetics of Anti-platelet Intervention" (PAPI) Study (NCT 00799396). Over a 6 week period participants will be given: 75 mg of clopidogrel for 8 days, at least 1 week washout, 150 mg of clopidogrel for eight days, at least 1 week washout, 300 mg of clopidogrel for eight days.
  Interventions: Drug: Clopidogrel
- Clopidogrel in extensive metabolizers (Experimental): Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI) will be recruited. We will select 6 extensive metabolizers (EM) to clopidogrel 75 mg from participants who previously received 75 mg clopidogrel as part of another NIH sponsored clinical trial entitled, "Pharmacogenetics of Anti-platelet Intervention" (PAPI) Study (NCT 00799396). Over a 6 week period participants will be given: 75 mg of clopidogrel for 8 days, at least 1 week washout, 150 mg of clopidogrel for eight days, at least 1 week washout, 300 mg of clopidogrel for eight days.
  Interventions: Drug: Clopidogrel
- Omeprazole/Clopidogrel in PM (Experimental): PM participants who have completed Arm 1 will have the option to participate. After a washout of at least one week, these participants will given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
  Interventions: Drug: Omeprazole/Clopidogrel
- Omeprazole/Clopidogrel in IM (Experimental): IM participants who have completed Arm 2 will have the option to participate. After a washout of at least one week, these participants will given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
  Interventions: Drug: Omeprazole/Clopidogrel
- Omeprazole/Clopidogrel in EM (Experimental): EM participants who have completed Arm 3 will have the option to participate. After a washout of at least one week, these participants will given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
  Interventions: Drug: Omeprazole/Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Over a 6 week period participants will be given: 75 mg of clopidogrel for 8 days, at least 1 week washout, 150 mg of clopidogrel for eight days, at least 1 week washout, 300 mg of clopidogrel for eight days.
  Other Names: Plavix
  Arms: Clopidogrel in extensive metabolizers; Clopidogrel in intermediate metabolizers; Clopidogrel in poor metabolizers
Drug: Omeprazole/Clopidogrel — After a washout of at least 1 week, participants will have the option to participate in a final intervention in which they will be given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
  Other Names: Prilosec; Plavix
  Arms: Omeprazole/Clopidogrel in EM; Omeprazole/Clopidogrel in IM; Omeprazole/Clopidogrel in PM

SUMMARY:
Clopidogrel (also known as Plavix) is used commonly in patients to prevent heart attacks and conditions caused by blood clots. Although clopidogrel works in many individuals, some people do not respond as well to this drug. The variation in treatment response may be linked to genetics. This study will examine the effects of clopidogrel in a population in which sequencing for certain genes has been performed in order to determine the role that genes play in the response to various clopidogrel maintenance doses.

DETAILED DESCRIPTION:
Clopidogrel is a prodrug with high inter-individual response variability. Clopidogrel is converted to an active drug in part through an enzyme encoded by the gene named CYP2C19. Individuals with genetically-impaired CYP2C19 metabolism have lower capacity to convert the prodrug to its active form. Consequently, these individuals have lower blood levels of the activated form of clopidogrel, diminished antiplatelet responses, and higher rates of cardiovascular events and stent thrombosis. Increasing doses of clopidogrel in such patients represents a possible approach to managing the gene-drug interaction.

The purpose of this study is to evaluate whether increasing the dose of clopidogrel increases antiplatelet responses and active metabolite exposure in individuals with genetically reduced CYP2C19 metabolism relative to those with normal CYP2C19 metabolism.

The primary objective is to assess changes in clopidogrel response and exposure at three clopidogrel dose levels and with coadministration of omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Amish men or women between 20 and 70 years of age who participated in PAPI

Exclusion Criteria:

* Severe hypertension (bp > 160/95 mm Hg)
* Co-existing malignancy
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 2 times normal
* Creatinine >2.0
* Hct < 32 or Hct > 50
* Thyroid Stimulating Hormone (TSH) < 0.40 or >5.50
* History of bleeding disorder or gastrointestinal bleeding
* History of unstable angina, myocardial infarction (MI), angioplasty, coronary artery bypass surgery
* History of atrial fibrillation, stroke or transient ischemic attacks or deep vein thrombosis
* Type 2 diabetes
* Thrombocytosis (platelet count > 500,000) or thrombocytopenia (platelet count < 150,000)
* Surgery within six months
* Clopidogrel allergy
* Pregnant women
* Currently breast feeding
* Omeprazole allergy
* Prospective participants taking medications that would affect the outcome(s) to be measured and who cannot willingly and safely, in the opinion of the treating physician and study physician, discontinue these medications for 1 week prior to protocol initiation, or who are taking vitamins and/or other supplements and who are unwilling to discontinue their use for at least 1 week prior to study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Horenstein, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Amish Research Clinic, Lancaster, Pennsylvania, United States

REFERENCES:
- [Background] Shuldiner AR, O'Connell JR, Bliden KP, Gandhi A, Ryan K, Horenstein RB, Damcott CM, Pakyz R, Tantry US, Gibson Q, Pollin TI, Post W, Parsa A, Mitchell BD, Faraday N, Herzog W, Gurbel PA. Association of cytochrome P450 2C19 genotype with the antiplatelet effect and clinical efficacy of clopidogrel therapy. JAMA. 2009 Aug 26;302(8):849-57. doi: 10.1001/jama.2009.1232. PMID 19706858
- [Background] Jiang XL, Samant S, Lewis JP, Horenstein RB, Shuldiner AR, Yerges-Armstrong LM, Peletier LA, Lesko LJ, Schmidt S. Development of a physiology-directed population pharmacokinetic and pharmacodynamic model for characterizing the impact of genetic and demographic factors on clopidogrel response in healthy adults. Eur J Pharm Sci. 2016 Jan 20;82:64-78. doi: 10.1016/j.ejps.2015.10.024. Epub 2015 Oct 30. PMID 26524713
- [Background] Horenstein RB, Madabushi R, Zineh I, Yerges-Armstrong LM, Peer CJ, Schuck RN, Figg WD, Shuldiner AR, Pacanowski MA. Effectiveness of clopidogrel dose escalation to normalize active metabolite exposure and antiplatelet effects in CYP2C19 poor metabolizers. J Clin Pharmacol. 2014 Aug;54(8):865-73. doi: 10.1002/jcph.293. Epub 2014 Apr 7. PMID 24710841

RESULTS

PARTICIPANT FLOW:
Groups:
- Poor Metabolizers: Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI (NCT00799396)) will be recruited. We will select 6 poor metabolizers to clopidogrel 75 mg from participants who previously received clopidogrel as part of another NIH sponsored clinical trial entitled, "Pharmacogenetics of Anti-platelet Intervention" (PAPI) Study (NCT00799396).
  Clopidogrel, Omeprazole: Over a 6 week period participants will be given:
  75mg of clopidogrel for 8 days, at least 1 week washout, 150mg of clopidogrel for eight days, at least 1 week washout, 300mg of clopidogrel for eight days. Participants will have the option to participate in a final week in which they will be given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
- Intermediate Metabolizers: Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI (NCT00799396)) will be recruited. We will select 6 intermediate metabolizers to clopidogrel 75 mg in PAPI (NCT00799396).
  Clopidogrel, Omeprazole: Over a 6 week period participants will be given:
  75mg of clopidogrel for 8 days, at least 1 week washout, 150mg of clopidogrel for eight days, at least 1 week washout, 300mg of clopidogrel for eight days. Participants will have the option to participate in a final week in which they will be given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
- Extensive Metabolizers: Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI (NCT00799396)) will be recruited. We will select 6 extensive metabolizers to clopidogrel 75 mg in PAPI (NCT00799396).
  Clopidogrel, Omeprazole: Over a 6 week period participants will be given:
  75mg of clopidogrel for 8 days, at least 1 week washout, 150mg of clopidogrel for eight days, at least 1 week washout, 300mg of clopidogrel for eight days. Participants will have the option to participate in a final week in which they will be given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
Period: Clopidogrel 75 mg
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Clopidogrel 150 mg
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Clopidogrel 225 mg
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Clopidogrel Plus Omeprazole
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Started | 5 | 5 | 4
Completed | 5 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Poor Metabolizers: Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI) will be recruited. We will select 6 poor metabolizers to clopidogrel 75 mg from participants who previously received clopidogrel as part of another NIH sponsored clinical trial entitled, "Pharmacogenetics of Anti-platelet Intervention" (PAPI) Study (NCT 00799396).
  Clopidogrel, Omeprazole: Over a 6 week period participants will be given:
  75mg of clopidogrel for 8 days, at least 1 week washout, 150mg of clopidogrel for eight days, at least 1 week washout, 300mg of clopidogrel for eight days. Participants will have the option to participate in a final week in which they will be given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
- Intermediate Metabolizers: Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI) will be recruited. We will select 6 intermediate metabolizers to clopidogrel 75 mg in PAPI (NCT 00799396).
  Clopidogrel, Omeprazole: Over a 6 week period participants will be given:
  75mg of clopidogrel for 8 days, at least 1 week washout, 150mg of clopidogrel for eight days, at least 1 week washout, 300mg of clopidogrel for eight days. Participants will have the option to participate in a final week in which they will be given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
- Extensive Metabolizers: Healthy subjects who have been genotyped for CYP2C19*2 and received clopidogrel as part of a prior study (PAPI) will be recruited. We will select 6 extensive metabolizers to clopidogrel 75 mg in PAPI (NCT 00799396).
  Clopidogrel, Omeprazole: Over a 6 week period participants will be given:
  75mg of clopidogrel for 8 days, at least 1 week washout, 150mg of clopidogrel for eight days, at least 1 week washout, 300mg of clopidogrel for eight days. Participants will have the option to participate in a final week in which they will be given 75 mg of clopidogrel together with 20 mg of omeprazole daily for eight days.
- Total: Total of all reporting groups
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 4 | 4 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Platelet Aggregation Following Therapy With Clopidogrel
Description: Adenosine diphosphate (ADP) mediated platelet aggregation measured 4 hours post-dose of clopidogrel on Day 1.
Time Frame: Day 1, 4 hours post clopidogrel dose
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Number analyzed (Participants) | 6 | 6 | 6
percentage of aggregation
  Clopidogrel 75mg | 62.9 (14.7) | 68.1 (5.0) | 62.5 (3.4)
  Clopidogrel 150mg | 63.2 (9.3) | 57.8 (7.2) | 53.9 (12.9)
  Clopidogrel 300mg | 53.3 (15.2) | 47.8 (13.6) | 38.6 (10.9)

2. Secondary Outcome: Change in Platelet Aggregation Following Therapy With Clopidogrel and Omeprazole
Description: The change in maximum platelet aggregation in response to ADP 4-hours post dose on day 8 of therapy with clopidogrel and omeprazole will be compared to the baseline measure of platelet aggregation at day 1 prior to drug therapy
Time Frame: Baseline, Day 8
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Number analyzed (Participants) | 5 | 5 | 4
percentage of aggregation | 11.6 (11.9) | 27.9 (9.3) | 37.5 (3.2)

3. Secondary Outcome: Level of Active Clopidogrel Metabolite
Description: The level of the active clopidogrel metabolite will be measured at at 0.25, 0.5, 1, 2, and 4 hours after the Day One dose is administered for pharmacokinetic analysis. The analysis will measure the Area Under the Curve.
Time Frame: Baseline, 0.25, 0.5, 1, 2, and 4 hours
Measure: Mean (Standard Deviation); unit: ng h/mL
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Number analyzed (Participants) | 6 | 6 | 6
ng h/mL
  Clopidogrel 75mg | 17.4 (19) | 33.3 (37) | 32.7 (25)
  Clopidogrel 150mg | 24.2 (26) | 43.8 (35) | 53.6 (35)
  Clopidogrel 300mg | 36 (35) | 73.7 (53) | 80.4 (24)

4. Primary Outcome: Change in Platelet Aggregation Following Therapy With Clopidogrel
Description: ADP mediated platelet aggregation measured 4 hours post Day 8 clopidogrel dose
Time Frame: 4 hours post Day 8 dose
Measure: Mean (Standard Deviation); unit: percentage of aggregation
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Number analyzed (Participants) | 6 | 6 | 6
percentage of aggregation
  Clopidogrel 75mg | 55.0 (14.5) | 37.8 (8.2) | 31.3 (7.3)
  Clopidogrel 150mg | 44.2 (15.0) | 33.2 (6.0) | 25.1 (7.1)
  Clopidogrel 300mg | 32.6 (10.7) | 25.7 (6.0) | 19.5 (6.9)

ADVERSE EVENTS:
Time Frame: Six weeks
Arm/Group | Poor Metabolizers | Intermediate Metabolizers | Extensive Metabolizers
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Poor Metabolizers (N=6) | Intermediate Metabolizers (N=6) | Extensive Metabolizers (N=6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — poison ivy
vasovagal reaction (Nervous system disorders) | 0 | 1 | 0
skin infection (Infections and infestations) | 0 | 0 | 1 — Fifths disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No